CLINICAL TRIAL: NCT07088601
Title: Efficacy of Oral Ondansetron Strips on Prevention of Post-Spinal Shivering; a Double Blinded, Randomized Controlled Study
Brief Title: Efficacy of Oral Ondansetron Strips on Prevention of Post-Spinal Shivering
Acronym: OOPS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hany Mohammed El-Hadi Shoukat Mohammed, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MS-442-2024
Record Dates: First submitted 2025-07-19; First posted 2025-07-28 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-12

CONDITIONS: Post-Spinal Shivering

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group O (Active Comparator): Patients will receive oral ondansetron in the form of an oral soluble film 4 mg strip.
  Interventions: Drug: Oral ondansetron strips
- Group C (Placebo Comparator): Patients will receive a placebo in the form of an oral peppermint strip
  Interventions: Other: Placebo (oral peppermint strip)

INTERVENTIONS:
Drug: Oral ondansetron strips — In the anesthesia preparation room and before the insertion of the peripheral IV cannula, patients in group O will receive oral ondansetron in the form of an oral soluble film 4 mg strip.
  Arms: Group O
Other: Placebo (oral peppermint strip) — In the anesthesia preparation room and before the insertion of the peripheral IV cannula, patients in group C will receive a placebo in the form of an oral peppermint strip.
  Arms: Group C

SUMMARY:
This study aims to investigate the efficacy of oral ondansetron film strips on the incidence of post-spinal shivering in patients undergoing surgeries using spinal anesthesia at Kasr Alainy hospitals, Cairo University.

This prospective, double-blinded, randomized controlled study will be conducted on 50 patients aged from 18 to 65 years of both sexes with ASA I, II who are scheduled for elective surgical procedures under spinal anesthesia in the lower half of the body such as orthopedic, urological, or general surgeries. Patients will be divided into two equal groups: Group (O) will receive oral ondansetron in the form of an oral soluble film 4 mg strip immediately before insertion of IV cannula and group (C) will receive a placebo in the form of an oral peppermint strip immediately before insertion of the IV cannula.

DETAILED DESCRIPTION:
In the anesthesia preparation room and before the insertion of the peripheral IV cannula, patients in group O will receive oral ondansetron in the form of an oral soluble film 4 mg strip (Ondalenz, 4 mg orodispersible films of Nerhadou International Co.) and patients in group C will receive a placebo in the form of an oral peppermint strip (Listerine Cool Mint Pocketpakas).

Following the insertion of a cannula; IV midazolam at a dose of 0.05 mg/kg will be administered intravenously. Then the patient will be transferred immediately to the operating theatre.

On entering the operating room; all patients will be connected to standard ASA monitoring which included electrocardiography (ECG), non-invasive arterial blood pressure (NIBP) including systolic, diastolic, mean arterial blood pressure (MAP) and Oxygen saturation using pulse oximetry.

With the patient sitting on the operating table, the L3-L4 interspace will be identified by identification of Tuffier's line. Under complete aseptic conditions, a dural puncture will be achieved by a 22G pencil-point spinal needle that will be introduced in a paramedian (lateral) approach through the L3-4 intervertebral space. After CSF aspiration and confirmation of correct intrathecal space, 3.5 mL of Sunny Pivacaine 0.5% (hyperbaric bupivacaine 20mg/4mL amp of Sunny pharmaceutical group) plus 25 μg of fentanyl-Hameln (of Sunny pharmaceutical group) will be injected over one minute.

The sensory block will be assessed by a pinprick test and the motor block will be assessed using a modified Bromage scale (0 = no motor block; 1= hip is blocked; 2= hip and knee are blocked; 3= hip, knee, and ankle are blocked). Peak sensory level will be confirmed and if a sensory level < T8 the patient will be excluded. If general anesthesia is needed for any reason, the patient will also be excluded from the study.

The ambient room temperature will be maintained at 24°C. IV fluids will be administered according to the conventional way as follows, hourly maintenance was the sum of A (4x first 10 Kg body weight), B (2x next 10 Kg body weight) and C (1x remaining Kg bodyweight) in addition to deficit (or fasting requirements), that will be hourly maintenance multiplied by the numbers of hours of fasting, half of it will be administered in the first hour and the second half will bne administered during second and third hours of surgery. Balanced crystalloids such as Ringer's lactate or acetate will be preferred over normal saline. Blood loss will be estimated through the surgical field, towels, gauzes and suction jar & will be replaced by crystalloids 1:3 or colloid/blood and blood products 1:1 ratio. All IV fluids will be administered at room temperature. All patients will be covered with surgical drapes from the lower extremities up to the lower chest during the operation. No warming devices will be used. Supplementary oxygen by a face mask will be given to all patients at a rate of 6 L/min.

The tympanic temperature will be monitored and measured by using the Braun ThermoScan 5 Ear Thermometer model IRT 6500. Hypothermia will be defined as a tympanic membrane temperature < 36.5◦ C.

Shivering score will then be assessed according to the Bedside shivering assessment score (BSAS) . If shivering scores ≥ 3, 30 mg of IV pethidine were administered as a rescue dose.

Postoperative:

Patients will be discharged to post anesthesia care unit (PACU). All patients will be monitored in the post-anesthesia care unit (PACU), covered by one cotton blanket over their entire body. The PACU temperature will be maintained at 24ºC.

The adverse effects will be assessed: allergic reaction from the used drugs, complications from the surgery done as:

Hypotension (MAP < 20% of baseline). In case of hypotension, the patients will be managed with intravenous loading with Ringer's lactate and boluses of 10 mg ephedrine IV.

Bradycardia (HR< 60 beats/min). In the case of bradycardia, the patients will be managed with 0.02 mg/kg atropine IV.

Respiratory depression will be considered if the respiratory rate is less than 10 breaths per minute and oxygen saturation (SpO2) was < 92% for 30 or more seconds.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I, II.
* Patients underwent elective surgical procedures under spinal anesthesia in the lower half of the body such as orthopedic, urological, or general surgeries.

Exclusion Criteria:

* Patient refusal.
* Morbid obese patients or those who were not candidates for spinal anesthesia.
* Pregnant females.
* Patients with comorbidities such as severe cardiopulmonary, severe hepatic or renal diseases, thyroid disorders, and convulsions.
* Uncooperative patients and patients with psychological disorders.
* Patients on regular ondansetron or other antiemetics.
* Patients taking selective serotonin reuptake inhibitors.
* Patients with allergy to 5-HT3 receptor antagonist drugs.
* Patients receiving saddle spinal block.
* In surgeries less than 1 h or longer than 3 hours duration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-10 (Estimated); Primary Completion 2025-12-29 (Estimated); Study Completion 2025-12-29 (Estimated)

PRIMARY OUTCOMES:
The incidence of shivering. | starting from 15 minutes after lumber puncture until 180 minutes following it and postoperative.
  It is defined by the highest shivering score ≥ 3 at any time starting from 15 min after lumber puncture until 180 min following it.

SECONDARY OUTCOMES:
The onset time of significant shivering | started from 15 minutes after lumbar injection until 180 minutes following lumbar injection and postoperative
  Time in min from the onset of significant shivering ≥ 3 on shivering score
Incidence of hypothermia | started from 15 minutes after lumbar injection until 180 minutes after lumbar injection and postoperative.
  Core body temperature will be measured by ear thermometer immediately before lumbar puncture (base level), and then at 15-minute intervals until 180 min after lumbar puncture and postoperative. Hypothermia will be defined as a tympanic membrane temperature < 36.5◦ C.
The shivering score | will be assessed at 15 minutes intervals during the operation and in the recovery room started from 15 minutes after the lumbar puncture until 180 minutes after the lumbar puncture and postoperative.
  Shivering score will be assessed according to the Bedside shivering assessment score (BSAS) as: Grade I: Mild fasciculation of face, neck, or head, or peripheral vasoconstriction, Grade II: Visible tremor involving one muscle group, Grade III Muscular activity in more than one muscle group but not generalized, and Grade IV: Gross muscular activity involving the entire body. The minimum is grade I and the maximum is Grade IV. Higher grades mean increased severity.
Incidence of patients given pethidine | started from 15 minutes after the lumbar puncture until 180 minutes after the lumbar puncture and postoperativde.
  If shivering scores ≥ 3, 30 mg of IV pethidine will be administered as a rescue dose.
Correlation between the incidence of shivering score ≥ 3 and hypothermia. | started 15 minutes after lumbar puncture until 180 minutes after lumbar puncture and postoperatively
  Correlation between the incidence of shivering score ≥ 3 as measured by Bedside Shivering Assessment Score (BSAS) and hypothermia as measured by tympanic thermometer (<36.5).
The incidence of adverse effects | started 15 minutes after lumbar puncture until 180 minutes after lumbar puncture and postoperatively
  e.g., hypotension, arrhythmias as bradycardia, nausea, vomiting, headache, itching, hypoxemia, and total spinal block) will be detected and recorded
Correlation between the incidences of postoperative nausea, vomiting, and shivering | started 15 minutes after lumbar puncture until 180 minutes after lumbar puncture and postoperatively

OTHER OUTCOMES:
Demographic data including age, sex, and weight | started immediately preoperatively until 1 minute before lumbar puncture
ASA physical status. | started immediately preoperatively until 1 minute before lumbar puncture
Heart rate | will be recorded at the following intervals: baseline (immediately before induction of spinal block), one minute after lumbar puncture, every 10 minutes in the first 30 minutes, then at 60 and 90 minutes intraoperatively and 30 minutes postoperatively
mean arterial blood pressure | will be recorded at the following intervals: baseline (immediately before induction of spinal block), one minute after lumbar puncture, every 10 minutes in the first 30 minutes, then at 60 and 90 minutes intraoperatively and 30 minutes postoperatively
oxygen saturation | will be recorded at the following intervals: baseline (immediately before induction of spinal block), one minute after lumbar puncture, every 10 minutes in the first 30 minutes, then at 60 and 90 minutes intraoperatively and 30 minutes postoperatively
respiratory rate | will be recorded at the following intervals: baseline (immediately before induction of spinal block), one minute after lumbar puncture, every 10 minutes in the first 30 minutes, then at 60 and 90 minutes intraoperatively and 30 minutes postoperatively